CLINICAL TRIAL: NCT06625086
Title: Investigation of the Effectiveness of a Web-Based Remote Exercise Program in Patients With Patellofemoral Pain Syndrome
Brief Title: Effect of Web-Based Exercise on Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-10840098-772.02-6172
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Rehabilitation; Telerehabilitation; Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Self-Guided Exercise Group (Active Comparator): A brochure explaining and demonstrating the exercises to be performed in treatment will be provided to 20 patients with PFPS. Patients will be asked to follow the exercise program for 6 weeks, 3 days per week, performing each exercise twice a day with 10 repetitions for each exercise.
  Interventions: Other: Convensional exercises
- Supervised Exercise Group (Experimental): Twenty patients with PFPS will perform exercises taught under the supervision of a physiotherapist for 6 weeks, 3 days per week, with each exercise performed twice a day and repeated 10 times.
  Interventions: Other: Supervised exercises
- Web-Based Exercise Group (Experimental): Group 3 (Web-Based Exercise Group): Twenty patients with PFPS will participate in a web-based exercise program for 6 weeks, 3 days per week, with each exercise performed twice a day and repeated 10 times.
  Web-Based Remote Exercise Program: The web-based application will be created using iOS and Android operating systems. Exercises specifically designed for PFPS treatment will be included in the application through video tutorials. Descriptive text explaining each exercise will be provided below each video. Information on how well each participant adheres to the exercise program, how frequently they perform each exercise, and their current status will be recorded.
  Interventions: Other: Web based exercises

INTERVENTIONS:
Other: Convensional exercises — Exercises will be provided to individuals in the Self-Guided Exercise group through a brochure.
  Arms: Self-Guided Exercise Group
Other: Supervised exercises — Exercises will be administered to individuals with PFPS under the supervision of a physiotherapist.
  Arms: Supervised Exercise Group
Other: Web based exercises — The exercises will be administered to participants through a web-based application.
  Arms: Web-Based Exercise Group

SUMMARY:
Patellofemoral pain syndrome (PFPS) is a common and challenging knee condition, characterized by pain around the patella. It primarily affects active women, athletes, and military personnel. PFPS accounts for a significant portion of musculoskeletal and knee complaints, though its true prevalence may be higher due to underdiagnosis. Diagnosis is based on a detailed history and physical exam, with symptoms like pain during activities such as kneeling, stair climbing, squatting, and running. The condition is caused by muscle imbalance, overactivity, overload, and trauma, leading to mechanical and dynamic control issues in the lower extremities.

Most PFPS treatments are conservative, focusing on physiotherapy approaches that include patient education, strengthening, flexibility, proprioception, and stretching exercises. Surgical interventions are rare.

Current literature lacks studies on the use of web-based remote exercise programs for PFPS patients. Therefore, this study aims to evaluate the effectiveness of a web-based, timed exercise program on pain, functional capacity, and kinesiophobia in individuals with PFPS.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is one of the most common and challenging knee disorders to treat. It refers to pain around the patella and surrounding structures. PFPS was first described in 1928 and is most frequently observed in active women, athletes, and military personnel. It accounts for a significant portion of musculoskeletal complaints and knee problems, and the actual prevalence may be higher as not all cases are diagnosed. The diagnosis of patellofemoral syndrome largely relies on a detailed and accurate history and physical examination. Symptoms can be unilateral or bilateral and often include pain associated with activities such as kneeling, stair climbing, squatting, and running. PFPS is characterized by an imbalance among the static and dynamic structures of the lower extremity, muscle imbalance, overactivity, overload, and trauma. Patients with PFPS exhibit abnormalities in mechanical and dynamic control of the lower extremity.

Most treatment approaches for PFPS are conservative, with surgical interventions being rare. Treatment programs typically involve a multimodal physiotherapy approach, including functional patient education, lower extremity strengthening, flexibility, proprioception, endurance, and stretching exercises.

Upon reviewing the existing literature, no studies were found that investigated the use of a web-based remote exercise program among patients with PFPS.

Therefore, the aim of this study is to investigate the effectiveness of a web-based remote, timed exercise program on pain, functional capacity, and kinesiophobia in individuals with patellofemoral pain syndrome. The evaluation will include the Visual Analog Scale (VAS) for pain assessment, the Tampa Scale for Kinesiophobia, the Kujala questionnaire for patellofemoral function, and the Timed Up and Go (TUG) test for functional mobility.

ELIGIBILITY:
Inclusion Criteria:

* Having atraumatic pain lasting for at least 3 months,
* Exhibiting characteristic signs of patellofemoral pain syndrome (retropatellar pain, the presence of the movie sign, and a positive patellar grind test),
* Having one or more positive patellofemoral pain triggers, such as prolonged sitting, squatting, kneeling, descending stairs, ascending stairs, or a positive patellar grind test,
* No knee instability and no grade 2-3 ligament or meniscus tears,
* Voluntary participation in the study.

Exclusion Criteria:

* A history of patellofemoral dislocation, subluxation, or osteoarthritis,
* A previous history of surgery or the presence of congenital deformity,
* The presence of neurological or rheumatological disease,
* Speech or comprehension impairment that affects communication,
* Having previously undergone physical therapy and rehabilitation for patellofemoral pain syndrome.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-10-05 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | From enrollment to the end of treatment at 6 weeks
  The Visual Analog Scale is used to measure the intensity of pain. The patient is asked to assess their pain on a line with values ranging from 0-10, where 0 means no pain, and 10 means unbearable pain. Individuals mark their pain intensity on this line according to their pain situation.
Kujala Patellofemoral Scoring | From enrollment to the end of treatment at 6 weeks
  The Kujala Patellofemoral Scoring scale was developed in 1993 by Kujala and colleagues to assess knee functionality in problems related to the patellofemoral structure. It has been proven to be a valid, reliable, and sensitive scale for patients with PFPS. The scale consists of 13 questions, and the scoring system ranges from 0 to 100, from worst to best. A higher score indicates better performance.
Time up and go test | From enrollment to the end of treatment at 6 weeks
  The Timed Up and Go (TUG) test is a functional assessment used to evaluate patients' mobility, balance, and walking abilities. Patients will be instructed to start from a seated position in a chair, stand up on command, walk as quickly as possible at a safe walking speed for a predetermined distance of 3 meters, turn around at the end point, and return to sit in the chair. The time from when they stand up until they sit down again will be recorded with a stopwatch. The test will be repeated three times, and the average time will be calculated.

SECONDARY OUTCOMES:
Tampa Scale for Kinesiophobia | From enrollment to the end of treatment at 6 weeks
  The Tampa Scale for Kinesiophobia, which has been validated for reliability in Turkish, will be used to assess kinesiophobia. The scale consists of 17 questions that inquire about avoidance of movement due to previous injury history or pain. The lowest score is 17, and the highest score is 68, with a score of 37 or above indicating a high level of kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

REFERENCES:
- [Derived] Menek B, Dansuk E. Comparative Efficacy of Supervised, Web-Based, and Self-Guided Exercise Interventions in Women with Patellofemoral Pain Syndrome. Medicina (Kaunas). 2025 Apr 15;61(4):731. doi: 10.3390/medicina61040731. PMID 40283022